CLINICAL TRIAL: NCT05636904
Title: A Proof-Of-Concept Phase 1b/2a Randomized, Vehicle, and Comparator-Controlled Study of Topical DLQ01 to Assess the Safety and Efficacy in the Treatment of Androgenetic Alopecia (AGA) in Men
Brief Title: Safety and Efficacy Study of Topical DLQ01 in the Treatment of Androgenetic Alopecia (AGA) in Men
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dermaliq Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DLQ01-001
Record Dates: First submitted 2022-11-16; First posted 2022-12-05 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia | interventions — Minoxidil; Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- DLQ01 high dose (Experimental): Twice daily application of DLQ01 high dose cutaneous solution in 30 subjects
  Interventions: Drug: prostaglandin F2a analogue in vehicle solution high dose
- DLQ01 low dose (Experimental): Twice daily application of DLQ01 low dose cutaneous solution in 30 subjects
  Interventions: Drug: prostaglandin F2a analogue in vehicle solution low dose
- active ingredient-free vehicle solution to DLQ01 (Placebo Comparator): Twice daily application of DLQ01 vehicle cutaneous solution in 30 subjects
  Interventions: Drug: active ingredient-free vehicle solution to DLQ01
- Minoxidil Solution 5% (Active Comparator): Twice daily application of the comparator cutaneous solution in 30 subjects
  Interventions: Drug: Minoxidil 5% Topical Solution

INTERVENTIONS:
Drug: prostaglandin F2a analogue in vehicle solution high dose — Topical treatment for 24 weeks
  Other Names: DLQ01 high dose
  Arms: DLQ01 high dose
Drug: prostaglandin F2a analogue in vehicle solution low dose — Topical treatment for 24 weeks
  Other Names: DLQ01 low dose
  Arms: DLQ01 low dose
Drug: active ingredient-free vehicle solution to DLQ01 — Topical treatment for 24 weeks
  Other Names: DLQ01 vehicle
  Arms: active ingredient-free vehicle solution to DLQ01
Drug: Minoxidil 5% Topical Solution — Topical treatment for 24 weeks
  Other Names: Regaine®
  Arms: Minoxidil Solution 5%

SUMMARY:
The goal of this study is to measure the safety, tolerability, and the hair growth response to topical DLQ01 solutions in comparison to the vehicle and a comparator solution in 120 males with Androgenetic Alopecia.

ELIGIBILITY:
Inclusion Criteria:

* Males with active AGA on the vertex area of the scalp consistent with Norwood-Hamilton Grades of IIIv through V, excluding IIIa, IVa, and Va grades.
* Willing to maintain the same hair style, approximate length, and hair colour throughout the duration of the study as documented in the global photograph at Day -2 of baseline.
* Willing to have target areas shaved and to have temporary dot tattoos placed on their scalp.
* Willing to comply with the study instructions and return to the site for required visits.
* Must be willing and able to communicate and participate in the entire study and willing to use an electronic diary to record investigational product dosing.
* Must provide written informed consent.

Exclusion Criteria:

* Participants with other type of alopecia other than AGA or any other concomitant skin or systemic disorder involving the scalp area.
* Participants with sensitive, irritated, or abraded scalp area.
* Participants who have undergone hair transplants or have had scalp reductions.
* Concurrent treatments or interventions that could affect interpretation of study data, prior to or during the study, as specified in the protocol
* Current evidence of another ongoing or acute relevant cutaneous infection, active systemic infection, or other significant skin conditions.
* History of relevant sensitivity to any of the study products, or components thereof, or a history of drug or other allergy that contraindicates study participation.
* Known allergy or sensitivity to tattoo ink.
* Participant with relevant active or prior history of malignancies.
* Participants with relevant cardiovascular disease including ischemic heart disease, cardiac arrhythmias, or congestive heart disease.
* History of any relevant alcoholism, substance or drug abuse-related disorders in the past year or a positive toxicology screening panel, or alcohol breath test at Screening.
* Clinically significant abnormal biochemistry, haematology or urinalysis values.
* Any other relevant serious illness or medical, physical, or psychiatric condition(s) that, could interfere with full participation in the study, pose a significant risk to the participant; or interfere with interpretation of study data.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
TAHC (total, terminal, and vellus) | 28 weeks
  Change from baseline in total, terminal, and vellus target area hair counts (TAHC) using digital image analysis after 4, 12, and 24 weeks of treatment, and at the follow-up visit
Cumulative hair thickness density (mm/cm2) | 28 weeks
  Change in cumulative hair thickness density using digital image analysis after 4, 12, and 24 weeks of treatment, and at the follow-up visit.
Anagen/telogen ratio | 28 weeks
  Change in anagen/telogen ratios using digital image analysis after 4, 12, and 24 weeks of treatment, and at the follow-up visit.

SECONDARY OUTCOMES:
Investigator global assessment (IGA) using a 7-point ordinal scale compared to baseline | 28 weeks
  Investigator assessment of the participant´s scalp hair growth compared to baseline using the following 7-point scale: greatly decreased (-3), moderately decreased (-2), slightly decreased (-1), no change (0), slightly increased (1), moderately increased (2), and greatly increased (3) compared to baseline at 4, 12, 16, and 24 weeks of treatment, and at the follow-up visit
Frequency of scores for cutaneous reactions in the treated area through study day 194 | 28 weeks
  Investigator assessment of cutaneous reactions such as erythema, oedema, glazing with fissures, vesicles, or papules, by grading with a clinical 5-point scale: no irritation (0), mild (1), moderate (2), severe (3), and very severe (4) at each visit through study day 194
Frequency of scores for pigmentation changes compared to non-treated area of scalp and hair through study day 194 | 28 weeks
  Investigator assessment of pigmentation changes compared to non-treated area of scalp and hair by grading with a clinical 4-point scale: no difference (0), slight difference, <25% (1), moderate difference, <50 to 75% (2), significantly darker/lighter, <75 to 100% (3) at each visit through study day 194
Number of participants with clinically significant abnormal laboratory test results | 28 weeks
  Collection of safety blood at screening, after 24 weeks of treatment, and at follow-up
Number of participants with clinically significant abnormal heart rate | 28 weeks
  Collection of heart rate at screening, baseline, and after 4, 16, and 24 weeks of treatment, and at follow-up
Number of participants with clinically significant abnormal blood pressure | 28 weeks
  Collection of blood pressure at screening, baseline, and after 4, 16, and 24 weeks of treatment, and at follow-up
Number of participants with clinically significant abnormal ECG readings | 28 weeks
  Collection of 12-lead ECG at screening, and after 4, 12, 16, and 24 weeks of treatment, and at follow-up
Plasma concentrations of DLQ01 | 24 weeks
  Blood samples for evaluation of plasma concentrations of active ingredient and novel excipient will be taken at baseline (predose) and after 4, 12 and 24 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Betsy Hughes-Formella, PhD, Study Director — Dermaliq Therapeutics, Inc.
Locations (2):
- Australia (2):
  - Dr Rodney Sinclair Pty Ltd,, East Melbourne, Victoria
  - Dr Rodney Sinclair Pty Ltd,, Pascoe Vale South, Victoria

IPD SHARING:
Plan to Share IPD: No